CLINICAL TRIAL: NCT01309516
Title: Efficacy of Learning Through Play Plus Intervention to Reduce Maternal Depression for Women With Under-nourished Children: A Randomized Controlled Trial From Pakistan
Brief Title: Randomised Control Trial of a Complex Intervention for Postnatal Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Dow University of Health Sciences (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pill110409
Record Dates: First submitted 2011-01-22; First posted 2011-03-07 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Postnatal Depression; Depression, Postpartum
Keywords: Postnatal depression; Maternal depression; Psychosocial intervention
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complex Intervention (LTP-TH) (Experimental): The 12 sessions of complex intervention (LTP-TH) will be delivered to mothers.
  Interventions: Behavioral: Complex Intervention
- Control group (No Intervention): Control group will receive standard postnatal follow-up.

INTERVENTIONS:
Behavioral: Complex Intervention — This 12 session Multimodal Psychosocial Intervention will include a supportive component, an educational component, psychosocial component and a parenting programme.
  Other Names: Multimodal Psychosocial Intervention
  Arms: Complex Intervention (LTP-TH)

SUMMARY:
The study aims to:

1. Develop a culturally appropriate psychosocial intervention
2. Test feasibility and acceptability of psychosocial intervention in women suffering from postnatal depression.

Primary Hypothesis:

Depressed mothers who will receive the group intervention will show significant improvements in terms of symptoms of depression.

Design:

Randomised controlled trial.

Setting:

Outpatient department of Civil hospital Karachi.

Participants:

A total of 84 depressed mothers will be randomised equally to an intervention group and a Treatment as usual control group.

Interventions:

The 12 session multimodal psychosocial intervention will be delivered to mothers in the intervention group over a three months period. Each session would take up to 45 minutes. Control group will receive standard postnatal follow-up.

Outcome measures:

Primary outcome measures would be mothers' scores on Edinburgh Postnatal Depression Scale (EPDS)and Hamilton Depression Rating Scale (HDRS).

DETAILED DESCRIPTION:
A number of individual and group interventions targeting maternal depression have been developed and tested, mostly in developed countries. Group-based approaches have usually been used to improve outcomes in children through parent-training programmes. A meta-analysis of such programmes shows that these can also be effective in improving psychosocial and mental health of the mothers. However, a number of health system and cultural differences make it difficult for mental health interventions to be extrapolated from the developed to the developing world.

Design:

The interventions will be assessed using a prospective randomised controlled design, using two groups: psychosocial group therapy (Learning Through Play + principles of Cognitive Behaviour Therapy)and treatment as usual.

Defining the intervention:

The intervention will include a supportive component, an educational component, and practical advice on using health services, a parenting component, and a psychosocial component. The objective will be to help mothers feel supported, empowered and confident about their parenting abilities, which in turn may help to reduce their level of depression. Further qualitative testing of the intervention will take place to refine the manualized intervention.

Psychiatric Measures:

The level of severity of depression will be assessed using the Edinburgh Postnatal Depression Scale (EPDS) (Cox and Holden, 1994) and the Hamilton Depression Rating Scale (HDRS) (Hamilton, 1960).

Women scoring 12 or over on the EPDS and 13 or over on the HDRS will be asked to undergo a diagnostic interview using the Clinical Interview Schedule-Revised (CIS-R).

To measure mother infant attachment the Maternal Attachment Inventory (Muller, 1994) will be used.

OSLO-3 item Social Support Scale (Dalgard, 1996) will be used to measure social support.

The adapted Verona Service Satisfaction Scale (Tansella, 1991) will be used to measure patient satisfaction with support and treatment.

Quality of life will be measured by using the EuroQol-5D (EQ-5D).

The qualitative interviews will be used to elicit information about previous attempts for help with mental health issues and questions regarding participants understanding of their postnatal depression and their future expectations from a perinatal service.

ELIGIBILITY:
Inclusion Criteria:

* Depressed mothers over the age of 18 years
* Having one or more infants 6-18 months old
* Ability to give informed consent
* Resident in the study catchment area

Exclusion Criteria:

* Women or child with diagnosed physical or learning disability and women having post-partum or other psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Depression | 6 months
  We will measure change from baseline in symptoms of depression through Hamilton Depression Rating Scale (HDRS) at six months by using 17 item HDRS.
Postnatal Depression | 6 months
  Edinburgh Postnatal Depression Scale (EPDS) will be used to identify mothers with postnatal depression.

SECONDARY OUTCOMES:
Infants' weight | 6 months
  Will be measured through standard anthropometric techniques and equipments
Infants' height | 6 months
  Will be measured through standard anthropometric techniques and equipments
Social Support | 6 months
  Social support of participants will be measured with OSLO 3-Items Social Support Scale
health related quality of life | 6 months
  EuroQol-5D(EQ-5 D) will be used to measures health related quality of life in five dimensions. It provides a simple descriptive profile and a single index value for health status.
Maternal Attachment | 6 months
  Maternal attachment with infants will be measured with Maternal Attachment Inventory (MAI)

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, MD, Principal Investigator — University of Manchester
Locations (2):
- Pakistan (2):
  - Civil hospital, Karachi, Sindh
  - Abbasi Shaheed hospital Karachi, Karachi, Sindh

REFERENCES:
- See also: Pakistan Institute of Learning & Living, Organization (Collaborator) offering logistic and technical support. — http://pill.org.pk